CLINICAL TRIAL: NCT00868075
Title: Pulmonary Rehabilitation in Non Cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Principal Investigator, Adam Hill, Consultant Physician and Honorary Senior Lecturer, NHS Lothian
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08/S1102/40
Record Dates: First submitted 2009-02-19; First posted 2009-03-24 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Bronchiectasis
Keywords: Physiotherapy; Rehabilitation; Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chest Physiotherapy (Experimental): Twice daily chest physiotherapy
  Interventions: Procedure: Chest physiotherapy
- Chest Physiotherapy + Exercise Program (Experimental): Chest Physiotherapy + Exercise Program
  Interventions: Procedure: Chest Physiotherapy + Exercise Program

INTERVENTIONS:
Procedure: Chest physiotherapy — Twice daily for 8 weeks
  Arms: Chest Physiotherapy
Procedure: Chest Physiotherapy + Exercise Program — Twice daily chest physiotherapy and Three times weekly exercise program (two sessions supervised)for 8 weeks
  Arms: Chest Physiotherapy + Exercise Program

SUMMARY:
The aim of our study is to ascertain whether chest physiotherapy + pulmonary rehabilitation is more efficacious than chest physiotherapy alone. The outcomes that will be used to assess effectiveness are relevant in terms of the direct benefit on the patient's health related quality of life.

PLANNED STUDY: This randomized study will compare 8 weeks chest physiotherapy with 8 weeks chest physiotherapy plus pulmonary rehabilitation.

DETAILED DESCRIPTION:
PLANNED STUDY: This randomized study will compare 8 weeks chest physiotherapy with 8 weeks chest physiotherapy plus pulmonary rehabilitation.

PLAN OF INVESTIGATION: Patients will be recruited from NHS Lothian with 15 randomized to chest physiotherapy and 15 to chest physiotherapy plus pulmonary rehabilitation.

Protocols:

Chest physiotherapy Physiotherapy will be aided using a positive pressure airways device (Acapella) that aids sputum expectoration. They will be asked to do 10 breaths, followed by 3 huffs and a cough. This will be repeated 3 times and repeated twice a day. Expected tiime 10-15 minutes twice daily.

Pulmonary rehabiliation Will be an 8-week programme twice a week in hospital with a third session (unsupervised) at home. It will include both cardiovascular training and upper limb and lower limb strengthening exercises.

Each patient will have a baseline exercise test. Calculation of the patient's 80% peak heart rate will be recorded and then used to ensure that patients are working to this level during the pulmonary rehabilitation cardiovascular sections.

The session will include: 5 minute warm up; 10 minutes treadmill; 10 minutes bicycle; 10 minutes stepper; 10 minutes upper limb and lower limb strengthening exercises; 5 minutes cool down.

Throughout the 8-week programme the resistance and intensity of each activity will be increased as they improve.

Following commencement of their first class they will be provided with a diary for a walking programme at home, which they will do once a week unsupervised.

Endpoints: Assessments below will be done at baseline, 4 weeks, 8 weeks and 3 months.

Microbiology: A fresh sputum sample will be submitted for micobiological culture.

Systemic inflammatory markers: 10mls venous blood for full blood count, erythrocyte sedimentation rate, C reactive protein, urea, electrolytes and liver function tests.

Pulmonary physiology: Pre bronchodilator spirometry (FEV1, FVC and FEV1/FVC), mouth pressures, followed by an incremental shuttle walk test.

24 hour sputum volume: This will be collected the day before each clinic visit. Sputum colour: Graded as mucoid, mucopurulent or purulent. Health related quality of life: Leicester Cough Questionnaire and St George's Respiratory Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate and severe bronchiectasis aged 18-75 will be recruited. Severity will be assessed radiologically by HRCT of the chest using the scoring method by Bhalla et al.

Exclusion Criteria:

* cystic fibrosis
* emphysema on HRCT chest and FEV1<60% predicted
* active allergic bronchopulmonary aspergillosis or tuberculosis
* poorly controlled asthma
* pregnancy or breast feeding
* current smokers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is improvement in exercise tolerance from an incremental walk test. | 8 weeks

SECONDARY OUTCOMES:
These include pulmonary physiology, 24 hour sputum volume, sputum appearance, health related quality of life and systemic inflammation. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adam T Hill, MD, FRCPE, Principal Investigator — NHS Lothian
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Derived] Mandal P, Sidhu MK, Kope L, Pollock W, Stevenson LM, Pentland JL, Turnbull K, Mac Quarrie S, Hill AT. A pilot study of pulmonary rehabilitation and chest physiotherapy versus chest physiotherapy alone in bronchiectasis. Respir Med. 2012 Dec;106(12):1647-54. doi: 10.1016/j.rmed.2012.08.004. Epub 2012 Sep 1. PMID 22947443